CLINICAL TRIAL: NCT02033720
Title: Neurological Outcomes After Cardiac Arrest in Pulseless Electrical Activity in Comparison to Asystole. Are All Non-shockable Rhythms the Same?
Brief Title: Study of Survivors of Different Types of Cardiac Arrest and Their Neurological Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Eyad AlThenayan, Dr. Eyad AlThenayan, University of Western Ontario, Canada
Other Study IDs: 104666
Record Dates: First submitted 2014-01-04; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Postcardiac Arrest; Pulseless Electrical Activity; Asystole
Keywords: postcardiac arrest; post cardiac arrest syndrome; post cardiac arrest hypothermia; pulseless electrical activity; asystole; therapeutic hypothermia; therapeutic hypothermia after cardiac arrest; therapeutic hypothermia neurologic outcome
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome | interventions — Hypothermia, Induced; Cool-Down Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Shockable arrest: Initial arrest rhythm shockable. This is either pulseless ventricular tachycardia (pulseless VT) or ventricular fibrillation (VF).
  Interventions: Other: No treatment; Other: Therapeutic hypothermia
- Pulseless electrical activity: Initial arrest rhythm is pulseless electrical activity.
  Interventions: Other: No treatment; Other: Therapeutic hypothermia
- Asystole: Initial arrest rhythm is asystole.
  Interventions: Other: No treatment; Other: Therapeutic hypothermia

INTERVENTIONS:
Other: No treatment — No therapeutic hypothermia was induced.
  Other Names: No therapeutic hypothermia.; Control.
Other: Therapeutic hypothermia — Hypothermia was induced after successful resuscitation from cardiac arrest.
  Other Names: Hypothermia; Induced hypothermia; Mild therapeutic hypothermia; Cooling; Targeted temperature management

SUMMARY:
After successful resuscitation from certain types of cardiac arrest, total body cooling is now a well established treatment that improves the chances of the brain recovering. This however, has only been definitively proven after a certain type of cardiac arrest that is "ventricular fibrillation / ventricular tachycardia". The purpose of this study is to explore if total body cooling is beneficial for patients recovering from another type of cardiac arrest that is "pulseless electrical activity".

HYPOTHESIS:

Patients undergoing post-cardiac arrest therapeutic hypothermia have better neurological outcomes if their initial arrest rhythm is pulseless electrical activity (PEA) in comparison to asystole.

DETAILED DESCRIPTION:
STUDY RATIONALE AND BACKGROUND INFORMATION:

After successful resuscitation from cardiac arrest the body experiences a period of global reperfusion. During this period, patients may show signs of myocardial stunning, lactic acidosis, neurological injury and reperfusion syndrome. This constellation of findings constitutes what is known as post-cardiac arrest syndrome. The brain appears to be one of the most vulnerable organs to injury during this reperfusion phase and varying degrees of cognitive impairment may be the end result. Inducing mild therapeutic hypothermia has been shown to be protective for the brain in this setting and has been demonstrated to improve neurological recovery. The evidence for this however, is only conclusive in cases where the arrest is in a shockable rhythm i.e. pulseless ventricular tachycardia and ventricular fibrillation.

In 2002, two randomized controlled trials were published showing an improvement in neurological outcomes in patients treated with mild therapeutic hypothermia post resuscitation from shockable cardiac arrest. Therapeutic hypothermia has since been widely adopted by most authorities as part of the comprehensive treatment bundle for post cardiac arrest syndrome. Whether there is any benefit for patients arrested in non-shockable rhythms however, is a matter of controversy. Some have reported improved mortality and better neurological outcomes with therapeutic hypothermia in this patient population. Others have reported no benefit or even a trend towards harm. And although the matter remains controversial, the recommendation still stands for therapeutic hypothermia to be offered for all comatose survivors of cardiac arrest whatever the arrest rhythm.

Most previous reports have examined the differences between shockable and non-shockable rhythms in terms of neurological outcome and mortality rates after therapeutic hypothermia. To our knowledge, no study has examined the differences in outcome between the two types of non-shockable rhythms, that is pulseless electrical activity (PEA) and asystole. We hypothesize that during PEA arrests, patients may retain some degree of cerebral perfusion and hence have better neurological outcomes post-resuscitation. That is in contrast to asystole where patients are likely to have no cerebral perfusion. In this study we attempt to detect any possible differences in neurological recovery (as indicated by the Cerebral Performance Category scale on hospital discharge) after therapeutic hypothermia, between patients arrested in PEA arrest and those arrested in asystole.

ELIGIBILITY:
Inclusion Criteria:

* Admission to adult ICU (age ≥18 years) at London Health Sciences Centre
* Primary reason for ICU admission: postcardiac arrest
* Both in-hospital and out-of-hospital cardiac arrest will be included
* ICU admission between Jan 2008 and Dec 2012.

Exclusion Criteria:

- ICU admissions primarily for reasons other than cardiac arrest.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care unit (ICU) with a diagnosis of postcardiac arrest between Jan 2008 and Dec 2012 will be examined.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Cerebral performance category score on hospital discharge | Upon discharge from hospital, assessed up to 36 months postcardiac arrest
  Neurological outcome on discharge from hospital as defined by the cerebral performance category (CPC) scale. The CPC scale is a 5 point scale. The outcome measure will be dichotomized into good or bad. Good outcome will be equivalent to CPC scores of 1 & 2 (where the patient is independent), and bad outcome will be equivalent to CPC scores of 3, 4 & 5 (where the patient is either dependent or dead).
  CPC Scale:
  1. Functioning normally and independent, possibly with a minor disability.
  2. Moderately disabled, still independent.
  3. Conscious but with a severe disability, dependent.
  4. Unconscious (comatose or in a persistent vegetative state).
  5. Brain dead or dead by traditional criteria.

SECONDARY OUTCOMES:
Hospital length of stay postcardiac arrest | Days spent in hospital after successful resuscitation from cardiac arrest, assessed up to 36 months from the date of cardiac arrest
  Hospital length of stay (LOS) post-cardiac arrest will be calculated from the day of the cardiac arrest to the day of hospital discharge. If prior to the arrest the patient was an inpatient, we will only count the days from the arrest to discharge. Days spent in hospital prior to the arrest will not be included.
Intensive care unit length of stay postcardiac arrest | Days spent in the intensive care unit after successful resuscitation from cardiac arrest, assessed up to 36 months from the date of cardiac arrest
  The length of stay (LOS) in the intensive care unit (ICU) in days, after successful resuscitation from cardiac arrest.
Neurological status after hospital discharge | Assessed up to 12 months from hospital discharge
  Neurological status as documented on the patient's first outpatient clinic visit, assessed up to 12 months from hospital discharge. This will be analyzed as a secondary outcome only if enough data is generated on chart review.

OTHER OUTCOMES:
Time to obeying commands | Assessed up to 21 days postcardiac arrest
  Total time in days from the cardiac arrest until the patient is able to obey commands, as documented in the patient's chart.
Documented negative neurological prognosticators | Upon withdrawal of life support, assessed up to 3 months postcardiac arrest
  For patient's in which the reason for withdrawal of life support is poor neurological outcome, the number of negative neurological prognosticators recorded in the chart will be examined.
  Examples of negative prognosticators include: negative somatosensory evoked potentials on post arrest day 3, post arrest status epilepticus, absent brain stem reflexes beyond post arrest day 2... etc.
Post arrest neurological investigations (including imaging studies) | Performed within 21 days from cardiac arrest
  All neurological investigations done within 21 days from cardiac arrest will be examined including electroencephalograms, somatosensory evoked potentials, brain magnetic resonance imaging, brain computerized tomography (CT) scans... etc.

CONTACTS AND LOCATIONS:
Overall Officials: Eyad Althenayan, MD, Principal Investigator — Western University, Canada; Philip Jones, MD, FRCPC, Study Director — Western University, Canada; Bryan Young, MD, FRCPC, Study Chair — Western University, Canada; Ahmed F Hegazy, MD, FRCPC, Study Director — Western University, Canada; Ana Igric, MD, FRCSC, Study Director — Western University, Canada; Carolyn Benson, MD, Study Director — Western University, Canada
Locations (2):
- Canada (2):
  - University Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario
  - Victoria Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario

REFERENCES:
- [Background] Holzer M. Targeted temperature management for comatose survivors of cardiac arrest. N Engl J Med. 2010 Sep 23;363(13):1256-64. doi: 10.1056/NEJMct1002402. No abstract available. PMID 20860507
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Hazinski MF, Nolan JP, Billi JE, Bottiger BW, Bossaert L, de Caen AR, Deakin CD, Drajer S, Eigel B, Hickey RW, Jacobs I, Kleinman ME, Kloeck W, Koster RW, Lim SH, Mancini ME, Montgomery WH, Morley PT, Morrison LJ, Nadkarni VM, O'Connor RE, Okada K, Perlman JM, Sayre MR, Shuster M, Soar J, Sunde K, Travers AH, Wyllie J, Zideman D. Part 1: Executive summary: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S250-75. doi: 10.1161/CIRCULATIONAHA.110.970897. No abstract available. PMID 20956249
- [Background] Arrich J; European Resuscitation Council Hypothermia After Cardiac Arrest Registry Study Group. Clinical application of mild therapeutic hypothermia after cardiac arrest. Crit Care Med. 2007 Apr;35(4):1041-7. doi: 10.1097/01.CCM.0000259383.48324.35. PMID 17334257
- [Background] Testori C, Sterz F, Behringer W, Haugk M, Uray T, Zeiner A, Janata A, Arrich J, Holzer M, Losert H. Mild therapeutic hypothermia is associated with favourable outcome in patients after cardiac arrest with non-shockable rhythms. Resuscitation. 2011 Sep;82(9):1162-7. doi: 10.1016/j.resuscitation.2011.05.022. Epub 2011 Jun 12. PMID 21705132
- [Background] Dumas F, Grimaldi D, Zuber B, Fichet J, Charpentier J, Pene F, Vivien B, Varenne O, Carli P, Jouven X, Empana JP, Cariou A. Is hypothermia after cardiac arrest effective in both shockable and nonshockable patients?: insights from a large registry. Circulation. 2011 Mar 1;123(8):877-86. doi: 10.1161/CIRCULATIONAHA.110.987347. Epub 2011 Feb 14. PMID 21321156